CLINICAL TRIAL: NCT00423241
Title: A Prospective, Randomized, Exploratory Comparison of the SEMPERFLO* Pain Management System to a Commercially Available Pain Relief System in Subjects Undergoing Open Inguinal Hernia Repair
Brief Title: SEMPERFLO* Pain Management System in Inguinal Hernia Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Market dynamics including other technologies made the project not viable.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Jonathan Batiller, MBA, Ethicon Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200-06-004
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Inguinal Hernia; Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEMPERFLO Pain Management System (Experimental)
  Interventions: Device: SEMPERFLO Pain Management System
- ON-Q PainBuster Post-Op Pain Relief System (Active Comparator)
  Interventions: Device: ON-Q PainBuster Post-Op Pain Relief System

INTERVENTIONS:
Device: SEMPERFLO Pain Management System — continuous infusion of 0.5% bupivacaine at 2mL per hour
  Other Names: Pain management system
  Arms: SEMPERFLO Pain Management System
Device: ON-Q PainBuster Post-Op Pain Relief System — continuous infusion of 0.5% bupivacaine at 2mL per hour
  Other Names: Pain management system
  Arms: ON-Q PainBuster Post-Op Pain Relief System

SUMMARY:
This study will compare the clinical performance of the SEMPERFLO* Pain Management System with another commercial pain relief system using 0.5% bupivacaine following unilateral, open, inguinal hernia repair procedures.

*Trademark

DETAILED DESCRIPTION:
Pain will be evaluated up to 5 days after surgery Subjects will be followed for 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a candidate for primary, non-emergent unilateral, open inguinal hernia repair procedure
* Subject is 18 years or older
* Subject must be willing to participate in the study, and provide informed consent to participate.

Exclusion Criteria:

* Subjects undergoing recurrent hernia repair;
* Subjects who plan to undergo another elective surgical procedure prior to the completion of this study;
* Subjects with known allergy to bupivacaine;
* Subjects with immunodeficiency diseases (including known HIV);
* Subjects with any findings identified by the surgeon that may preclude conduct of the study;
* Subjects who are known current alcohol and/or drug abusers;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Dynamic pain (pain measured with coughing) measured using a ten-point visual analog scale | twenty-four hours post procedure

SECONDARY OUTCOMES:
Narcotic and non-narcotic analgesic usage | 24, 48, 72, 96 and 120 hours post- procedure
Numeric pain scale scores at rest and with coughing | 24, 48, 72, 96, and 120 hours post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (6):
- United States (6):
  - Boca Raton Community Hospital, Boca Raton, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Washington University, St Louis, Missouri
  - Universtiy of Tennessee, Knoxville, Tennessee
  - North Texas Surgery Center, Dallas, Texas
  - Michale E. DeBakey VA Medical Center, Houston, Texas